CLINICAL TRIAL: NCT05349513
Title: Interest of the Tool: Evaluation of Specific Care in an Ecological Environment for Patients Suffering From Schizophrenia-like Disorders
Acronym: IEvaEcoSchi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022-A00080-43
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Patients With Schizophrenia-like Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventionnal arm (Experimental): Administration of the experimental questionnaire ESSME in patient's environment.
  Interventions: Other: ESSME questionnaire

INTERVENTIONS:
Other: ESSME questionnaire — The experimental ecological questionnaire ESSME is administered 7 to 14 days after the inclusion visit and 7 to 14 days after the 6 months follow-up visit to the patient at their home.

SUMMARY:
The study use a new ecological questionnaire called ESSME developed by a care team in order to evaluate ecological environment of patients with schizophrenia-like disorders.

Indeed, evaluation in an ecological environment would make it possible to be as close as possible to the concerns of theses patients, which could improve the care of this population, by making it possible to set with the patient objectives anchored in their daily life.

DETAILED DESCRIPTION:
The duration of patient's participation to the study is 6 months plus 7 to 14 days.

The study includes the following visits :

* V0: Inclusion visit (Day 0) with the administration of standard of care questionnaires;
* V1: visit at patient's home (Day 0 +7 to 14 days) with the administration of the experimental ESSME questionnaire;
* V2: follow-up visit at 6 months (M6) with the administration of the same standard of care questionnaires than at the inclusion visit;
* V3: visit at patient's home (M6 + 7 to 14 days) with the administration of the experimental ESSME questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* man or woman aged 18 to 65 inclusive;
* diagnosis of schizophrenia or schizoaffective disorder according to the Diagnostic and Statistical Manual of Mental Disorders version number 5 (DSM-V) criteria;
* patient receiving care in a Center for Rehabilitation and Intersectoral Therapeutic Activities (CREATIV);
* person who consented to the study;
* affiliate or beneficiary of a social security scheme.

Exclusion Criteria:

* patient aged under 18 or over 65;
* pregnant or breastfeeding women;
* person unable or unwilling to receive a home visit;
* person not consenting to the study;
* presence of a diagnosis of an associated neurodevelopmental disorder;
* presence of a diagnosis of dementia or associated neurodegenerative process;
* person with a level of French language insufficient to understand the items.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between the total ecological questionnaire (ESSME) score and the total score of the social autonomy scale. | 6 months
  The main judgment criterion is the correlation coefficient between the change in the total ESSME score and the change in the total score of the selected autonomy scale, the EAS over a period of 6 months.
  The judgment criterion will be obtained by calculating a percentage variation between the initial total score and that obtained at 6 months for each of the scales: EAS and for the ESSME tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Henri Laborit, Poitiers, France

IPD SHARING:
Plan to Share IPD: No